CLINICAL TRIAL: NCT06157151
Title: A Randomized, Open-label, Two-arm, Multicenter Phase 2 Study to Evaluate Efficacy and Safety of PRGN-2009 in Combination With Pembrolizumab Versus Pembrolizumab Monotherapy in Patients With Recurrent or Metastatic Cervical Cancer.
Brief Title: PRGN-2009 in Combination With Pembrolizumab Versus Pembrolizumab in Patients With Recurrent or Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Precigen, Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRGN-2009-201
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer; HPV-Related Carcinoma; HPV-Related Malignancy; Recurrent Cervical Carcinoma; Metastatic Cervical Cancer
Keywords: Human Papilloma Virus; Cervical Cancer; Pembrolizumab; Therapeutic Vaccine; Cervix Cancer; Resistance to Checkpoint Inhibitors
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRGN-2009 plus Pembrolizumab (Experimental): PRGN-2009 at a dose of 5 x 10^11 PU q3W for 3 administrations, then q6w, plus Pembrolizumab, 400mg q6w
  Interventions: Biological: PRGN-2009 plus Pembrolizumab
- Pembrolizumab alone (Active Comparator): Pembrolizumab, 400mg q6w
  Interventions: Drug: Pembrolizumab alone

INTERVENTIONS:
Biological: PRGN-2009 plus Pembrolizumab — Subjects randomized will receive PRGN-2009 (5 x 10^11 PU, subcutaneous (SC) injection) every 3 weeks for three administrations, thereafter subjects will continue to receive PRGN-2009 administrations every 6 weeks. Pembrolizumab will be administered concurrently as intravenous (IV) infusion (400 mg) every 6 weeks.
  Arms: PRGN-2009 plus Pembrolizumab
Drug: Pembrolizumab alone — Subjects randomized will receive IV infusion of pembrolizumab (400 mg) administered every 6 weeks.
  Arms: Pembrolizumab alone

SUMMARY:
This randomized trial will evaluate the efficacy and safety of PRGN-2009 in combination with pembrolizumab compared to pembrolizumab alone in patients with pembrolizumab-resistant recurrent or metastatic cervical cancer.

DETAILED DESCRIPTION:
This is a randomized, two-arm study of PRGN-2009 in patients with recurrent or metastatic cervical cancer who are pembrolizumab resistant. Patients meeting all eligibility criteria who consent to participate in the study will be randomized 1:1 to receive a combination of PRGN-2009, plus pembrolizumab, or to receive pembrolizumab alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Recurrent or metastatic cervical cancer (histologically or cytologically confirmed) that meets the criteria of pembrolizumab-resistant.
* Must have been treated with pembrolizumab, either as monotherapy or in combination
* Patients must have received no more than two prior systemic regimens in the recurrent or metastatic setting
* Tumors are confirmed positive for PD-L1 and HPV16/18
* Measurable disease that can be accurately measured by RECIST v1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥ 12 weeks from the time of enrollment.
* Must have adequate organ function
* Negative serum pregnancy test. Women of child-bearing potential (WOCBP) must agree to use adequate contraception prior to study entry and for at least 6 months following completion of study treatment.
* All patients must have the ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Patients with presence of other active malignancy within 1 year prior to study entry
* Known Central Nervous System (CNS) disease
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Known history of active tuberculosis (TB, Bacillus tuberculosis).
* Pregnant and lactating women are excluded from this study.
* Patients with a history of solid organ transplant.
* Patients currently participating in a study of an investigational agent or have used an investigational device within 4 weeks prior to the first dose of study treatment.
* Patients, who in the opinion of the investigator, may not be able to comply with the monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Determine the Objective Response Rate (ORR) following treatment with PRGN-2009 in combination with pembrolizumab or pembrolizumab alone in patients with pembrolizumab-resistant recurrent or metastatic cervical cancer. | 1 year
  The ORR will be calculated as the combination of subjects achieving a complete response or a partial response per RECIST v1.1.
  ORR will be calculated and presented with 2-sided 95% confidence interval.

SECONDARY OUTCOMES:
Safety of PRGN-2009 in combination with pembrolizumab or pembrolizumab alone | 1 year
  Systemic toxicity will be assessed through the capture of Treatment Emergent Adverse Events ( TEAEs). The severity of the TEAEs will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 scale.
Progression-Free Survival (PFS) and Overall Survival (OS) following treatment with PRGN-2009 in combination with pembrolizumab or pembrolizumab alone | 1 year
  Duration of PFS and OS will be summarized using the Kaplan-Meier Product Limit estimator along with the corresponding two sided-95% Confidence intervals.
Best Overall Responses (BOR) and Disease Control Rate (DCR) per RECIST v1.1 following treatment with PRGN-2009 in combination with pembrolizumab or pembrolizumab alone | 1 year
  The proportion of subjects with BOR and DCR will be summarized using descriptive statistics.
Time to Response and Duration of Responses following treatment with PRGN-2009 in combination with pembrolizumab or pembrolizumab alone | 1 year
  TTR and DOR will be summarized using descriptive statistics.
Vector shedding following subcutaneous administration of PRGN-2009 | Up to 4 months
  Samples collected before and at specific intervals after treatment will be evaluated for presence of adenoviral vector.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - National Institute of Health, Bethesda, Maryland
  - University of Washington, Seattle, Washington